CLINICAL TRIAL: NCT05380986
Title: A Real World Study of Camrelizumab Combined With Apatinib Mesylate in Solid Tumors
Brief Title: Camrelizumab Combined With Apatinib Mesylate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, LiNing, Associate Chief Physician, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-RWS
Record Dates: First submitted 2022-05-10; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Solid Tumor
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab combined with apatinib mesylate (Experimental): Camrelizumab 200 mg, IVGTT D1, apatinib mesylate, once daily. The specific prescription is determined by the investigator. Continued use until disease progression, unacceptable toxicity, or withdrawal for other reasons.
  Interventions: Drug: Camrelizumab combined with apatinib mesylate

INTERVENTIONS:
Drug: Camrelizumab combined with apatinib mesylate — Camrelizumab 200 mg, IVGTT D1, apatinib mesylate, once daily. The specific prescription is determined by the investigator. Continued use until disease progression, unacceptable toxicity, or withdrawal for other reasons.

SUMMARY:
The purpose of this study is to observe the safety of camrelizumab combined with apatinib mesylate in the treatment of solid tumors

DETAILED DESCRIPTION:
According to current studies, the combination of camrelizide and apatinib mesylate has significant efficacy and controllable toxicity in the treatment of solid tumors.

This study adopted camrelizumab combined with apatinib mesylate in the treatment of solid tumors, aiming to further explore the safety of camrelizumab combined with apatinib mesylate in the treatment of solid tumors and provide more research data for the treatment of solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years old, male or female;
2. ECOG score is 0~2;
3. Patients with solid tumors confirmed by pathology or histology;
4. At least one measurable lesion (according to RECIST V 1.1);
5. For patients who have failed first-line or second-line treatment or who cannot tolerate standard treatment regimens for solid tumors.
6. Estimated survival ≥3 months;
7. Patients who have used immunosuppressants or antiangiogenic drugs in the past are not excluded;
8. For women who have not undergone menopause or surgical sterilization, agree to abstain from sex or use an effective contraceptive method during treatment and for at least 7 months after the last dose given in study treatment;
9. Researchers think they can benefit;
10. Voluntarily participate in the study and sign the informed consent;

Exclusion Criteria:

1. Pregnant or lactating women;
2. Except patients with contraindications to camrelizumab and/or apatinib mesylate, that is, those allergic to camrelizumab and its excipients; Allergic to apatinib mesylate should be prohibited; It should be contraindication for patients with active bleeding, ulcers, intestinal perforation, intestinal obstruction, hypertension beyond drug control within 30 days after major surgery, class III-IV cardiac insufficiency (NYHA standard), and severe hepatic or renal insufficiency (Class 4).
3. Those deemed unsuitable for inclusion by doctors;
4. The researchers determined there was a high risk that the tumor would invade important blood vessels and cause fatal hemorrhages during the follow-up study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-05-20 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
AE | up to 2 years
  any adverse medical event that occurs after a subject or clinical study receives a drug or treatment regimen

SECONDARY OUTCOMES:
Objective response rate | up to 2 years
  Defined as the proportion of patients with a documented complete response, and partial response (CR+PR)
Disease control rate | up to 2 years
  defined as the proportion of patients with complete response, partial response and disease stabilization (CR+PR+SD)
Overall survival | up to 2 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Tumor Hospital, Henan, China